CLINICAL TRIAL: NCT05833282
Title: Prognostic Factors and Therapeutic Management of ESBL Enterobacteriaceae in the ICU
Acronym: BLSE-REA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tourcoing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NRIPH_2023_01
Record Dates: First submitted 2023-04-04; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Drug Resistance, Multiple, Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multicenter retrospective study conducted in the intensive care units of Tourcoing, Roubaix, and Lille hospitals. Patients hospitalized in the ICU with EBLSE bacteremia within 24 hours before or during their stay in the ICU will be selected from microbiology laboratory data. Patient demographics and clinical data will be collected from the medical record. Microbiological results will be collected from the laboratory data.

DETAILED DESCRIPTION:
INCLUSION CRITERIA - Patients admitted to the ICU with EBLSE bacteremia within 24 hours before or during their stay in the ICU.

PRIMARY ENDPOINT

- The primary endpoint is 30-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU with EBLSE bacteremia within 24 hours before or during their stay in the ICU.

Exclusion Criteria:

* Patient who is a minor, protected adult, or who refuses to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU with EBLSE bacteremia
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is all-cause 30-day mortality. | 30-day mortality
  all-cause mortality.

SECONDARY OUTCOMES:
Adequacy of initial antibiotic therapy to french recommendations | adequate within 30 days
  Antibiotic prescriptions will be considered adequate if all of the following criteria meet the recommendations: molecule, dose, according to the recommendations provided by the French Society of Infectious Diseases. The recommendations for prescribing antibiotics are similar to those proposed by international guidelines.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier DRON, Tourcoing, France

IPD SHARING:
Plan to Share IPD: Undecided